CLINICAL TRIAL: NCT06262503
Title: The Influence of Virtual Reality Approach on Phantom Pain in Trans Tibial Amputation: A Randomized Control Trail
Brief Title: the Influence of Virtual Reality Approach on Phantom Pain in Trans Tibial Amputation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Medhat Helal Mohamed, physiotherapy partctitioner, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004810
Record Dates: First submitted 2024-02-08; First posted 2024-02-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Phantom Pain Following Amputation of Lower Limb
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Group1:conventional physiotherapy for phantom Pain Group2:conventional physiotherapy and Virtual Reality for phantom Pain
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1(Control ) (Other): Will receive conventional physiotherapy for one month and measure the pain intensity and lower extremity function
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS); Device: Mirroring Therapy; Other: Phantom Exercises
- Group2 (Experimental) (Experimental): Will receive conventional physiotherapy and Virtual Reality for phantom Pain for one month and measure the pain intensity and lower extremity function
  Interventions: Device: Virtual Reality; Device: Transcutaneous Electrical Nerve Stimulation (TENS); Device: Mirroring Therapy; Other: Phantom Exercises

INTERVENTIONS:
Device: Virtual Reality — Virtual Reality device is used for creating 3d avatar to engage the patient into a virtual world so he can overcome his pain
  Arms: Group2 (Experimental)
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — TENS stimulation plays on pain gate theory it sends stimulation to close C-fibers to relieve the pain and make the patient comfortable. The electrodes were put around the stump leg (residual limb) and the session lasts for 15 minutes, the parameters were Conventional TENS - high frequency (50-100 Hz), low intensity, short pulse width (50-200 μs). Pain relief by means of the pain gate mechanism involves activation (excitation) of the A beta (Aβ) sensory fibers, and by doing so, reduces the transmission of the noxious stimulus from the 'c' fibers, through the spinal cord and hence on to the higher centers.
Device: Mirroring Therapy — Mirroring Therapy :it tricks the brain. By placing a mirror between the healthy limb and the missing limb, patients see a reflection of the healthy limb, essentially "replacing" the phantom limb with a visual representation. This visual feedback is thought to reactivate brain areas responsible for the missing limb, potentially restoring its representation and reducing the discomfort of PLP. Essentially it aims to heal the brain's image of the body, which might in turn alleviate the pain associated with the missing limb.
Other: Phantom Exercises — The study investigated phantom exercises (PE) for phantom limb pain (PLP) relief. Patients performed specific foot and leg movements 15 times, stopping if PLP disappeared early. Exercises were repeated daily or upon PLP recurrence. Patients imagined their phantom limb position and mimicked it with their remaining limb, performing ankle, foot, knee, and hip movements until relaxation and PLP subsided.

SUMMARY:
1. To investigate the effect of Virtual reality (VR) on phantom limb pain in trans tibial amputation.
2. To investigate the effect of Virtual reality (VR) on lower limb Function in trans tibial amputation.

A sample size of 60 will be randomly allocated to two groups(30 in each group) , by using computer-generated random number list method. Control group will receive conventional physiotherapy(TENS- Phantom exercises and mirroring exercise) for reducing phantom pain in trans -tibial amputation and the experimental group will receive conventional physiotherapy(TENS- Phantom exercises and mirroring exercise) and Virtual Reality for reducing phantom pain in trans -tibial amputation .

DETAILED DESCRIPTION:
Pain management has become an increasingly important healthcare concern in clinical practice.

The investigators use the phrase (phantom nerve pain) for pain described by patients related to the absence of sensation. Though simple numbness is often well-tolerated and not bothersome, phantom nerve pain develops for some patients.

The painful area is essentially numb yet painful, hence the term "anesthesia dolorosa," which translates as "painfully numb." In a similar way to amputees who have phantom limb pain (PLP) in a limb no longer present, patients with peripheral nerve injury can have phantom nerve pain in the denervated area. The investigators hypothesize that damage to the peripheral first-order neurons, along with spontaneously firing second-order neurons, causes this pain and, if not treated in a timely manner, results in cortical remodeling and centrally mediated pain (as in phantom limb pain).

Phantom limb pain (PLP) is experienced by 65-85% of limb amputees. In addition, a range of other sensations can originate in the missing limb including phantom limb awareness, phantom sensations (such as itching and pins and needles), and kinetic and kinesthetic sensations (movement and position in space). Traditionally the treatment target has been PLP; however, it has become clear over many years that treatment options have limited success.

Although in many cases these phenomena do not cause suffering, phantom limb- distortions often co-occur with phantom limb pain (PLP) , in other words, a painful sensation located in the phantom and thus outside the physical borders of the body. PLP is reported by the majority of amputees , accounts for a significant reduction in health-related quality of life and only insufficiently responds to conventional pharmacological interventions The large variation in symptomatology suggests a multifactorial origin of phantom phenomena. It has been shown that the amputation induces negative effects on peripheral and central physiological mechanisms, both contributing to the experience of phantom phenomena including PLP.

The two most common types of Lower limb Amputation (LLAs) are transfemoral amputation (TFA) and trans-tibial amputation (TTA). TFAs make up 31% of all amputations, and TTAs make up 39% of all amputations .

Virtual Reality (VR) is characterized by an artificial computer-generated environment created to replace real-world sensory inputs ,It uses a computer to generate a simulation environment, which the users interact with, providing an immersive experience that facilitates the perception of being physically present in the virtual environment. In recent years, with the advent of more affordable devices such as head-mounted displays, VR has become a more feasible and popular technology ). Unlike many analgesics, which disrupt the C-fiber pathway that relays nociceptive signals to the central nervous system, VR affects pain perception through attention, concentration, and emotional alteration.( The immersive environment created by VR reduces pain experience by up-regulating nonpainful neural signaling. Increasing evidence supports VR as an alternative strategy for acute, burn, and experimental pain management in both adults and children. Additional experiments have demonstrated the positive effect of VR on pain in a variety of medical procedures including chemotherapy and wound care.

With immersive technology, participants view the full panorama, which enables the creation of a high sense of presence and immersion as if the participant is essentially inside the created environment.

One of the strategies for the management of PLP is phantom motor execution (PME), also known as phantom exercises. PME involves the imaginary movement of phantom limb in the brain along with the performance of certain actual physical movements. Neurophysiological networking involved in PME is similar to that of actual executed physical activities of sound limb and it should be distinguished from pure imaginary activities as it follows a different neurophysiological pathway . Such exercises have been shown to safely and effectively relieve PLP in various types of limb amputations .

ELIGIBILITY:
Inclusion Criteria:

1. All participants were prescreened older than 18 years; able to provide informed consent; with unilateral traumatic Factors Phantom Limb Pain lower limb amputation after complete recovery.
2. chronic PLP for more than 3 months.
3. If the subject was taking any medications, dosages must have been stable for at least 2 weeks before enrollment in the study.
4. Normal Body mass index ranged from 18.5 to 24.9.

Exclusion Criteria:

1. History of alcohol or drug abuse within the past 6 months.
2. Medical history of photophobia, epilepsy or any other light sensitivity.
3. Visual impairment thought to render the test invalid (people who need to wear glasses day to day are not excluded.
4. Uncontrolled epilepsy or prior seizures within the past year.
5. History of unexplained fainting spells or loss of consciousness as self-reported during the past 2 years.
6. Mirror therapy within 3 months prior to enrollment.

Ages: 18 Months to 75 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity Level | 4 weeks
  Pain Intensity Level is measured by McGill Pain Questionnaire to determine the pain level The McGill Pain Questionnaire. The descriptors fall into four major groups: sensory (S)1-10, affective (A) 11-15, evaluative (E), 16 and miscellaneous (M)17-20. The rank value for each descriptor is based on its position in the word set. The sum of the rank values is the pain rating index (PRI). The present pain intensity (PPI) is based on a scale of (0-5) 0 refers to no pain and 5 refers to worst pain and know the effectiveness of the Virtual Reality wither pain is increased or decreased .
Lower Extremity Functional | 4 weeks
  Lower Extremity Functional is measured by Lower Extremity Functional Scale (LEFS) to know the progress of patient movement and balance.It is divided to 5 categories; 0 indicates extreme difficult or unable to perform activity, 1 indicates quite a bit of difficulty, 2 indicates moderate difficulty, 3 indicates a little bit of difficulty, 4 indicates no difficulty

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical therapy, Cairo university, Giza, Egypt